CLINICAL TRIAL: NCT05495165
Title: Feasibility of Early Nutritional Prehabilitation Through a Therapeutic Education Programme for Cancer People With Potential Risk of Malnutrition
Brief Title: Early Education Programme in Malnourished Cancer Patients
Acronym: NEHOTEL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beauvais Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: NEHOTEL
Record Dates: First submitted 2022-05-17; First posted 2022-08-10 (Actual); Last update posted 2022-08-12 (Actual); Status verified 2022-08

CONDITIONS: Nutrition Aspect of Cancer
Keywords: Malnutrition; cancer; prehabilitation; therapeutic education
MeSH Terms: conditions — Malnutrition; Neoplasms | interventions — Nutritional Status; Psychology

STUDY DESIGN:
Intervention Model Description: 60 patients entered a 5-day educational device and then followed monthly for 8 months remotely by a smart phone application and dietary consultations.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nutritional educative programme (Other): 5 days educative programme before treatment
  Interventions: Other: Therapeutic education for patients in nutrition

INTERVENTIONS:
Other: Therapeutic education for patients in nutrition — Stakeholders give preventive therapeutic education recommandations in their specific expertize
  Other Names: Therapeutic education for patients in sophrology; Therapeutic education for patients in socio-aesthetic; Therapeutic education for patients in adapted physical activity; Therapeutic education for patients in psychology

SUMMARY:
The innovation is based on the proposal to integrate the patient, just after the announcement, before or at the beginning of the treatment (before the third session of chemotherapy or radiotherapy), in a 5-day training course in a clinical site that inspires peace of mind involving the family caregiver. The therapeutic education programme is led by a multidisciplinary team whose approach is centred on dietetics, supported by tools for encouragement via socio-aesthetics, physical activity and sophrology.

The educational objective is to promote the autonomy of the patient as well as the family caregiver, to involve them in the care pathway alongside the practitioners, with a view to contain undernutrition and reverse the spiral that increases the risks of morbi-mortality.

The aim of the study is to assess patient adherence to the device, the technical and economic feasibility, and its impact on quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* From 18 to 70 years old
* Patient with an ORL, pancreatic, oesogastric, duodenal or broncho-pulmonary cancer
* Patient who have not begun their treatments or patient in the beginning of their treatments, less than or equal to two sessions of chemotherapy or radiotherapy
* patient living in a private home (personal or family)
* Prognosis greater than 12 months
* Decision taken at a multidisciplinary consultation meeting (RCP) for a curative treatment
* WHO Score Performance Status ≤2
* Patient undernourished at the advertisement codes E44.1 "Mild protein-energy malnutrition" or E44.0 "Moderate protein-energy malnutrition", according to the latest HAS recommendations
* Patient not undernourished at the time of the announcement, but going to receive a treatment or combination of treatments for curative purposes, whose therapeutic sequences are known to induce nutritional complications inducing a risk of stopping treatment
* Per os nutrition
* With internet access and reachable by phone
* Patient affiliated to the social security system
* Patient information and signature of informed consent
* Patient accompanied by a family member or not

Exclusion Criteria:

* Patient with severe malnutrition corresponding to at least one of the criteria* below:

  (i) BMI < 17 kg/m². (ii) weight loss ≥ 10% in 1 month or ≥ 15% in 6 months or ≥ 15% of the usual weight before the onset of the disease (iii) albuminemia ≤ 30 g/L. (*) Annex 15.8: HAS 2019 source : A single criterion of severe undernutrition takes precedence over one or more criteria of moderate undernutrition.
* Treatment for curative purposes not applicable
* Comorbidities that do not allow participation in the prehabilitation course (patient presenting at least one of the criteria below):

Weight greater than 130kgs (limit of resistance of the beds in the reception centre) Sensory deficits: visual, auditory, olfactory, gustatory (not allowing to follow the educational workshops) Cognitive deficit (reading, writing, counting) Physical (ability to move around and participate in activities) Patient at risk of alcohol withdrawal

* TNM coupled with a deteriorated general condition of the patient at the time of the announcement; prediction of highly mutilating surgery involving an inability to eat through the mouth; metastatic stage.
* Patient institutionalized and/or not responsible for his or her diet
* Patient requiring parenteral or artificial enteral nutrition (feeding tube, nasogastric tube, gastrostomy or feeding jejunostomy)
* History of organ failure (cirrhosis, moderate or severe renal failure, heart failure (NYHA>2), chronic oxygen-dependent respiratory failure)
* Anaemic patient (hemoglobin level less than 9g/dL)
* Person deprived of liberty or under guardianship
* Inability to undergo the medical monitoring of the trial for geographical, social or psychological reasons.
* Pregnant woman or Breastfeeding woman
* A delay before the first treatment does not allow inclusion in the NEHOTEL prehabilitation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Rate of acceptance | during the 5-days programme
  Evaluation of the rate of screening failures and the explanation of refusals when the program is offered to patients (CONSORT Standards)
Rate of patients' skills development during the therapeutic educative programme | 8 months
  Rate of patients completing the stay and demonstrating ongoing or effective acquisition on 18 skills (self-reported questionnaire and confronted with observations of nursing staff) (acquired, in progress of acquisition, not acquired)
Programme and environment (hosting) satisfaction questionnaire assessment | during the 5-days programme
  Patient's motivational level during the therapeutic educative programme
Acceptance of treatment assessment | 8 months
  Alliance to care during the 8 months of follow-up via the IDP. This is measured by the number of PTE sessions the patients enroll and by questions on the application of the nutritional advices given during the intervention week
Assessment of the programme's cost | during the 5-days programme
  Calculation of "cost-utility" and "cost-effectiveness" based on a group of 6 people by PTE session
Real cost estimation | during the 5-days programme
  Estimation of avoided costs and calculation of the difference with the actual consolidated cost of the NEHOTEL stay

SECONDARY OUTCOMES:
Quality of Life Questionnaire related to cancer (QLQ C30) to assess the patients' quality of life | 8 months
  Scale from 0 (worse quality of life) to 100 (best quality of life)
Quality of Life Questionnaire Head and Neck (QLQ H&N35) to assess the patients' quality of life | 8 months
  Scale from 0 (worse quality of life) to 100 (best quality of life)
Number of therapeutic events completed | 8 months
  Number of therapeutic events completed compared to the initial objective (IDP)
The count of adverse events related or not to treatment | 8 months
  The count of adverse events related or not to treatment
Anthropomorphic markers (weight in kilograms) | 8 months
  Evolution of cancer biomarkers (IDP) to asses the evolution of undernutrition
Anthropomorphic markers (height in meters) | 8 months
  Evolution of cancer biomarkers (IDP) to asses the evolution of undernutrition
anthropomorphic markers (weight and height are used to calculate the BMI in kg/m^2) | 8 months
  evolution of cancer biomarkers (IDP) to asses the evolution of undernutrition
Biological markers (quantity of albumine in blood) | 8 months
  Evolution of cancer biomarkers (IDP) to asses the evolution of undernutrition
Biological markers (quantity of lymphocyte in blood) | 8 months
  Evolution of cancer biomarkers (IDP) to asses the evolution of undernutrition
Biological markers (quantity of albumine and lymphocyte in blood are used to calculate the PNI with the formula [10 * taux albumine (g/dL)] + [nombre de lymphocytes totaux/µL * 0,05]) | 8 months
  Evolution of cancer biomarkers (IDP) to asses the evolution of undernutrition
Food intake quantity and quality estimation with the Visual Analogue Scale (VAS) | 8 months
  Scale from 0 (no food intake) to 10 (normal quatity food intake) to assess the evolution of undernutrition
Consumption of Nutritional Oral Complements (NOC) | 8 months
  Evolution of NOC's consumption to assess the evolution of undernutrition
Borg Rating Scale of Perceived Exertion (Borg) scale after a physical activity to assess the physical activity and the effectiveness of reinforcement tools | 8 months
  Score between 0 (no perceived effort) and 20 (perceived effort maximal)
International Physical Activity Questionnaire (IPAQ) to assess the physical activity and the effectiveness of reinforcement tools | 8 months
  Evolution of the time of intense activity, moderate activity, light intensity and sedentary
World Health Organisation (WHO) scale to evaluate the capacity to move to assess the physical activity and the effectiveness of reinforcement tools | 8 months
  Scale from 0 (same capacity than before the surgery) to 4 (incapacity to move alone)
Drawing test Questionnaire to assess the socio-aesthetic programme and the patients' self-esteem | 8 months
  Evolution between the first drawing test at the beginning of the week and the second at the end
Rosenberg Self-Esteem Scale (Rosenberg) questionnaire to assess the socio-aesthetic programme and the patients' self-esteem | 8 months
  Final score between 10 (worse self-esteem and 40 (best self-esteem))
Hospital Anxiety and Depression (HAD) scale to assess the sophrology programme and the patients' anxiety and depression | 8 months
  Two scales (one for anxiety and one for depression) from 0 (worse well-being) to 21 (best well-being)
European Quality of Life-5 Dimensions Visual Analogue Scale (EQ-5D-VAS) to assess the sophrology programme and the patients' well-being | 8 months
  Scale from 0 (worse health) to 100 (best health)

OTHER OUTCOMES:
Zarit scale to evaluate the motivation and the effectiveness of the presence of the caregiver | during the 5-days programme
  Scale from 0 (taking care is not constraining for the caregiver) to 88 (taking care is a very heavy load for the caregiver)
Getting started with the eCRF application (Diétis) by patients | during the 5-days programme
  Rate of errors in filling in the Dietis tool by patients during the intervention week.
  Number of times the Dietis tool questionnaires were completed by patients during the intervention week
Assessment of the level of adherence to the application tool (Diétis) during the follow-up of 8 months | 8 months
  Rate of complete questionnaires and responses to the dietétician calls during the follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Sif Dr Bendjaballah, Doctor, Principal Investigator — Beauvais Hospital

IPD SHARING:
Plan to Share IPD: No
The PNI will be calculated by the following equation: [(10 × serum albumin (g/dL)) + (0.005 × total lymphocyte count)].
  Albumin Pre-albumin CRP Haemoglobin

REFERENCES:
- [Background] Arends J, Bachmann P, Baracos V, Barthelemy N, Bertz H, Bozzetti F, Fearon K, Hutterer E, Isenring E, Kaasa S, Krznaric Z, Laird B, Larsson M, Laviano A, Muhlebach S, Muscaritoli M, Oldervoll L, Ravasco P, Solheim T, Strasser F, de van der Schueren M, Preiser JC. ESPEN guidelines on nutrition in cancer patients. Clin Nutr. 2017 Feb;36(1):11-48. doi: 10.1016/j.clnu.2016.07.015. Epub 2016 Aug 6. PMID 27637832